CLINICAL TRIAL: NCT00839891
Title: A Phase 1 Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel Group/Crossover Thorough QT/QTc Study to Evaluate the Effect of a Therapeutic Dose and a Supra-therapeutic Dose of VI-0521 on Cardiac Repolarization in Healthy Male and Female Volunteers
Brief Title: A Study to Evaluate How VI-0521 Affect Cardiac Repolarization in Healthy Male and Female Volunteers
Acronym: TQT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, VP Clinical, Vivus, inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: OB-118
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2010-01

CONDITIONS: Torsades de Pointes
Keywords: TQT, QTc
MeSH Terms: conditions — Torsades de Pointes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3 (Placebo Comparator): Group 1: 56 subjects to receive active study drug (VI-0521) at steady state, PHEN/TPM 7.5/46 (a potential therapeutic dose), escalating to PHEN/TPM 22.5/138 (a supra-therapeutic dose);
  Group 2: 28 subjects to receive placebo preceded by a single oral dose of moxifloxacin on Day 2;
  Group 3: 28 subjects to receive placebo followed by a single oral dose of moxifloxacin on Day 24;
  Interventions: Drug: VI-0521

INTERVENTIONS:
Drug: VI-0521 — PHEN/TPM 7.5/46 mg (a potential therapeutic dose) PHEN/TPM 22.5/138 mg (a supra-therapeutic dose)

SUMMARY:
* Determine whether VI-0521 has an effect on the electrical activity of the heart in healthy subjects.
* Find out how much VI-0521 is in the blood and any potential side effects on ECG's of healthy subjects after taking the study drugs.

DETAILED DESCRIPTION:
This three-arm, parallel group, double-blind, active- and placebo-controlled study comparing VI-0521 at a potential therapeutic dose of PHEN/TPM 7.5/46 and PHEN/TPM 22.5/138 , a supra-therapeutic dose, with placebo. A single oral dose of 400 mg moxifloxacin is included as a positive control in terms of the effect on cardiac repolarization. The three treatment regimens are defined as follows:

Group 1: 56 subjects to receive active study drug (VI-0521) at steady state, PHEN/TPM 7.5/46 (a potential therapeutic dose), escalating to PHEN/TPM 22.5/138 (a supra-therapeutic dose);

Group 2: 28 subjects to receive placebo preceded by a single oral dose of moxifloxacin on Day 2;

Group 3: 28 subjects to receive placebo followed by a single oral dose of moxifloxacin on Day 24;

A total of 112 healthy subjects (with an approximate 1:1 female:male ratio) are planned to be randomized.Subjects will check into the clinical research unit (CRU) on Day -1. Day 1 will be a baseline electrocardiogram (ECG) profile day (all groups). Active dosing for Group 1 with VI-0521 will commence on Day 2. VI-0521 dose will escalate every 2-3 days until steady-state is achieved on Day 10 for the therapeutic dose PHEN/TPM 7.5/46. A full ECG assessment day will be performed (all groups, blinded); enabling the comparison of VI 0521 PHEN/TPM 7.5/46 with the placebo (pooled Groups 2 and 3).Subsequently, VI-0521 doses will be escalated until subjects in Group 1 reach a dose of 22.5/138, and then continue at this dose level until Day 22. On Day 22, when the active group has reached a steady state for the supratherapeutic dose level, another ECG assessment day will be performed (all groups, blinded); enabling a comparison of supratherapeutic VI-0521 with placebo (pooled Groups 2 and 3). Groups 2 and 3 will receive VI-0521 placebo on Days 2 to 22.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged 19 to 50 years, inclusive.
* Body mass index (BMI) between 24 and 30 kg/m2, inclusive.
* Subjects must be in good health, as determined by a medical history, physical examination, 12-lead ECG and clinical laboratory evaluations.
* Women of child-bearing potential should test negative for pregnancy, must use medically acceptable contraceptive methods

Exclusion Criteria:

* Male subjects with a resting QTcB or QTcF value <320 msec or >450 msec, and female subjects with a resting QTcB or QTcF value <320 msec or >470 msec, as measured at the screening visit.
* Subjects with clinically significant ECG abnormalities that may interfere with the accurate assessment of the QT interval, including intraventricular conduction delays (QRS >120 msec) and complete bundle branch blocks.
* Subjects who have a history of, or risk factors for, Torsades de Pointes (TdP) (eg, heart failure, abnormal serum electrolytes), including a family history of arrhythmia, sudden death or long QT syndrome.
* Subjects with known clinically significant arrhythmias or rhythm disturbances observed on the screening ECG and confirmed by a subsequent 24-hour ECG Holter recording.
* Subjects who have a supine heart rate (HR) at screening outside 45 to 90 beats per minute (bpm) (measured following at least a 10-minute rest).
* Subjects suffering from, or with a history of, one or more of the following conditions: hypertension, impaired glucose tolerance, diabetes mellitus, renal disease, edema, stroke or neurological disorder, rheumatological disorder (including arthritis, joint or tendon abnormalities), pulmonary disorder (including personal history of asthma), cardiovascular disorder (including coronary heart disease, congestive heart failure, cardiomyopathy, and any valvular heart disease), hepatic disorder, or a history of any illness that, in the opinion of the Investigator, might confound the results of the study or pose additional risk to the subject by participation in the study.
* Subjects with a history of psychiatric disorders, including bipolar disorder, psychosis, previous episode(s) of major depression or current depression, history of suicidality or suicidal ideation.
* Subjects with a history of nephrolithiasis or cholelithiasis.
* Subjects with a history of glaucoma, increased intraocular pressure, or use of any medication to treat increased intraocular pressure.
* Laboratory values at screening that are outside the normal range for the site unless prior approval is obtained from the VIVUS, Inc. medical monitor or designee.
* Subjects who are currently regular users (including recreational use) of any illicit drugs or who have a history of drug (including alcohol) abuse within 1 year of screening.
* Subjects who drink excessive amounts (equivalent to >4 cups of brewed coffee per day) of coffee, tea, cola or other caffeinated beverages within the 2 weeks prior to Day -1.
* Subjects with a positive urine drug test at screening and/or on Day -1 (eg, cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids).
* Subjects who consume excessive amounts of alcohol, defined as >3 drinks (beer, wine or distilled spirits) of alcoholic beverages per day, have a history of alcohol abuse, or are unwilling to comply with the restricted use of alcohol during the study.
* Subjects with a positive test for ethanol at screening and/or on Day -1.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess whether treatment with a potential therapeutic dose or a supra-therapeutic dose of VI-0521 has the potential to cause QT/QTc prolongation in healthy volunteers. | 25 days

SECONDARY OUTCOMES:
A secondary objective is to demonstrate assay sensitivity by showing that the active control (moxifloxacin 400 mg) treatment, corrected for placebo, produces a QTc change >5 msec. | 25 Days

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, PhD, Study Director — Clinical Pharmacology Consultant
Locations (1):
- MDS Pharma Services, Phoenix, Arizona, United States